CLINICAL TRIAL: NCT01228539
Title: Breaking the Cycle IV: Military PTSD (MPTSD) Treatment Study
Acronym: MPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Julian Ford, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPTSD-10-118-2; DOJ-2009-D1BX0299 (Other Grant/Funding Number: National Institute of Justice, Department of Justice)
Record Dates: First submitted 2010-09-22; First posted 2010-10-26 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: PTSD; Anger; Aggression
Keywords: PTSD; Anger; Aggression; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TARGET (Experimental): Affect regulation psychotherapy for PTSD
  Interventions: Behavioral: TARGET (Trauma Affect Regulation)
- Prolonged Exposure (Active Comparator): Cognitive behavioral therapy for PTSD with trauma memory exposure
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: TARGET (Trauma Affect Regulation) — TARGET teaches a skill sequence for affect regulation and social/interpersonal information processing.
  Other Names: TARGET
  Arms: TARGET
Behavioral: Prolonged Exposure — Cognitive behavior therapy with trauma memory exposure
  Arms: Prolonged Exposure

SUMMARY:
The study will compare the efficacy of Trauma Affect Regulation: Guide for Education and Therapy (TARGET) vs. the best validated psychotherapy for adults with posttraumatic stress disorder (PTSD), Prolonged Exposure (PE). Male military personnel and veterans suffering with PTSD and problems with anger after returning from military service in Afghanistan (Operation Emerging Freedom, OEF) and/or Iraq (Operation Iraqi Freedom, OIF) will be participants. The goal is to determine if a present-centered psychotherapy that teaches skills for emotion regulation and does not require re-telling of traumatic memories is as efficacious as the trauma memory-focused PE psychotherapy.

DETAILED DESCRIPTION:
The study is based on a theoretical and clinical model that involves a series of associated risks that are set in motion by exposure to military-related traumatic stressors in Iraq or Afghanistan. Trauma exposure places personnel at risk for PTSD, which in turn increases their risk of problems with anger and hostility, emotion dysregulation and experiential avoidance, and ultimately with alcohol abuse and aggression. The two types of treatments being compared, TARGET (Trauma Affect Regulation: Guide for Education and Therapy) and PE (Prolonged Exposure), are both designed to directly reduce PTSD severity by reducing emotion dysregulation (TARGET) and experiential avoidance (PE), and therefore are hypothesized to reduce the risk and severity of alcohol abuse and aggression- and thereby to reduce associated legal and societal costs.

ELIGIBILITY:
Inclusion Criteria:

* be a returning OEF/OIF military personnel or veteran
* have experienced PTSD for the past month
* have experienced anger and at least one act of aggression in the last month
* be mentally able to provide a valid consent

Exclusion Criteria:

* currently be danger of suicide
* currently abusing alcohol or other substances
* been in an inpatient psychiatric or addiction treatment program in the past month

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Severity of PTSD symptoms | Post-therapy
  Clinician Administered PTSD Scale Ordinal Scores Posttraumatic Cognitions Inventory Trauma Memory Questionnaire Interpretation of PTSD Symptoms Scale

SECONDARY OUTCOMES:
Anger/aggression problems | Post-therapy
  State-Trait Anger Expression Inventory Brief Symptom Inventory
Emotion Regulation | Post-therapy
  Negative Mood Regulation scale Difficulty with Emotion Regulation Scale Acceptance and Action Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Julian Ford, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States